CLINICAL TRIAL: NCT05128773
Title: A Randomized, Multicenter, Double-blind, Phase 3 Study of Amcenestrant (SAR439859) Versus Tamoxifen for the Treatment of Patients With Hormone Receptor-positive, Human Epidermal Growth Factor Receptor 2-negative or Positive, Stage IIB-III Breast Cancer Who Have Discontinued Adjuvant Aromatase Inhibitor Therapy Due to Treatment-related Toxicity
Brief Title: Study of Amcenestrant (SAR439859) Versus Tamoxifen for Patients With Hormone Receptor-positive (HR+) Early Breast Cancer, Who Have Discontinued Adjuvant Aromatase Inhibitor Therapy Due to Treatment-related Toxicity
Acronym: AMEERA-6
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern
Sponsor: Sanofi (Industry)
Collaborators: Breast International Group (Other); Alliance Foundation Trials, LLC. (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16133; U1111-1244-1767 (Registry Identifier: ICTRP); BIG 20-01 (Other: BIG); AFT-55 (Other: AFT); EORTC-2033 (Other: EORTC); 2021-000398-10 (EudraCT Number)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amcenestrant with tamoxifen-matching placebo arm (Experimental): Amcenestrant dose, once daily, continuously. Tamoxifen-matching placebo, once daily, continuously.
  Interventions: Drug: Amcenestrant; Drug: Tamoxifen-matching placebo
- Tamoxifen with amcenestrant-matching placebo (Active Comparator): Tamoxifen dose, once daily, continuously. Amcenestrant-matching placebo, once daily, continuously.
  Interventions: Drug: Tamoxifen; Drug: Amcenestrant-matching placebo

INTERVENTIONS:
Drug: Amcenestrant — tablet, oral
  Arms: Amcenestrant with tamoxifen-matching placebo arm
Drug: Tamoxifen — tablet, oral
  Arms: Tamoxifen with amcenestrant-matching placebo
Drug: Amcenestrant-matching placebo — tablet, oral
  Arms: Tamoxifen with amcenestrant-matching placebo
Drug: Tamoxifen-matching placebo — tablet, oral
  Arms: Amcenestrant with tamoxifen-matching placebo arm

SUMMARY:
This was a phase III, randomized, double blind, multicenter, 2-arm study evaluating the efficacy and safety of amcenestrant compared with tamoxifen in participants with hormone receptor-positive early breast cancer who discontinued adjuvant aromatase inhibitor (AI) therapy due to treatment related toxicity. The primary objective was to demonstrate the superiority of amcenestrant versus tamoxifen on invasive breast cancer-free survival.

The treatment duration per participant was to be 5 years, followed with a subsequent 5-years follow-up period. For the treatment period, visits were scheduled at the start of treatment, then at 4 weeks and 12 weeks after treatment start, and then every 12 weeks for the first 2 years and every 24 weeks for year 3 to 5. For the follow-up period, visits were scheduled 30 days after last treatment and then every 12 months. Three periods were planned:

* A screening period of up to 28 days,
* A treatment period of up to 5 years,
* A follow-up period of up to 5 years.

DETAILED DESCRIPTION:
Study duration per participant was to be approximately 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with histologically confirmed diagnosis of adenocarcinoma of the breast with documentation of hormone receptor-positive status, irrespective of human epidermal growth factor receptor 2 (HER2) status NOTE: Participants with HER2-positive breast cancer were eligible only if they had completed their adjuvant anti-HER2 treatment and chemotherapy.
* With Stage IIB or Stage III (invasive breast cancer) who had undergone breast surgery and adjuvant radiation (if indicated) for the current malignancy.
* Who had received prior aromatase inhibitors (AIs) (letrozole, anastrozole or exemestane or any sequence thereof) per the following:

Adjuvant AI therapy was discontinued due to AI treatment-related toxicity; Minimum of 6 months duration and maximum of 30 months duration (from initiation of first AI if there was a switch between AIs) of AI therapy was required.

* Absence of locoregional and/or advanced/metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Capable of giving signed informed consent.

Exclusion Criteria:

* Medical history or ongoing gastrointestinal disorders potentially affecting the absorption of amcenestrant and/or tamoxifen. Participants unable to swallow normally or unable to take tablets and capsules. Predictable poor compliance to oral treatment. Active inflammatory bowel disease or chronic diarrhea, active hepatitis A/B/C, hepatic cirrhosis, short bowel syndrome, or any upper gastrointestinal surgery including gastric resection or banding procedures.
* History of prior breast cancer treated with AI.
* Any other solid tumor or lymphoma diagnosis was not allowed except if the participant had been free from disease for equal to greater than (=>5) years.
* Pregnant or nursing women, or women of child-bearing potential without a negative pregnancy test prior to randomization.
* Participants with unrecovered acute toxic effects of prior AI therapy or surgical procedures.
* Uncontrolled intercurrent illness, including psychiatric conditions that would have limited compliance with study requirements.
* Treatment with any selective estrogen receptor degrader (SERD), tamoxifen or toremifene were not allowed as prior adjuvant therapy but could have been used as neoadjuvant therapy for a total duration of 3 months. Participants who were treated with a SERD, tamoxifen or toremifene in the neoadjuvant setting and who experienced disease progression were not allowed. Prior treatment with raloxifene or tamoxifen for bone health, risk reduction, or a prior breast cancer was allowed provided this was discontinued at least 3 years before diagnosis of current breast cancer.
* Ongoing treatment with HER2 directed therapy. Appropriate wash out between the last dose of HER2 directed therapy and randomization should have been at least 4 weeks.

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Brain, MD PhD, Study Chair — Institut Curie (Saint-Cloud and Paris), 35 rue Dailly, 92210 Saint-Cloud; David Cameron, Professor of Oncology, Study Chair — University of Edinburgh Cancer Centre, institute of Genetics and Cancer, Western General Hospital, Crewe Road South, EDINBURGH EH4 2XU Scotland; Otto Metzger, MD, Study Chair — Dana-Farber Cancer Institute, 450 Brookline Avenue Yawkey 1250
Locations (2):
- Investigational Site Number :1521622, Santiago, Reg Metropolitana de Santiago, Chile
- Investigational Site Number :1561599, Haikou, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16133 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25240&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 active centers in Chile and China. A total of 6 participants were screened between 17 February 2022 and 11 August 2022, of which 3 participants were randomized and exposed to study treatment.
Pre-assignment Details: Randomization stratified by prior exposure to (neo)adjuvant aromatase inhibitor therapy, (neo)adjuvant chemotherapy & HER2 status, CDK4/6 inhibitor (Yes/No), geographic regions, men' or peri-/pre-menopausal women vs. post-menopausal women. Study was initially planned with two treatment arms (i.e. amcenestrant & tamoxifen), however no participants were exposed to tamoxifen arm due to premature discontinuation & study closure by sponsor thus none of the participants were enrolled in tamoxifen arm.
Groups:
- Amcenestrant 200 mg + Tamoxifen-Matching Placebo: Participants received amcenestrant 200 mg along with tamoxifen-matching placebo orally (PO), once a day (QD) from Day 1 to Day 28 of each 28-day treatment cycle and were followed-up until diagnosis of disease recurrence per invasive breast cancer-free survival (IBCFS) definition (recurrence of one of following: Ipsilateral invasive breast tumor recurrence (IIBTR); local-regional invasive breast cancer recurrence; distant recurrence, invasive contralateral breast cancer, death) or any other withdrawal criterion whichever occurs first (maximum exposure duration: 155 days).
Period: Overall Study
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Started | 3
Completed | 0
Not Completed | 3
Not completed — Sponsor decision to terminate study | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the randomized population.
Groups:
- Amcenestrant 200 mg + Tamoxifen-Matching Placebo: Participants received amcenestrant 200 mg along with tamoxifen-matching placebo orally PO, QD from Day 1 to Day 28 of each 28-day treatment cycle and were followed-up until diagnosis of disease recurrence per IBCFS definition (recurrence of one of following: IIBTR; local-regional invasive breast cancer recurrence; distant recurrence, invasive contralateral breast cancer, death) or any other withdrawal criterion whichever occurs first (maximum exposure duration: 155 days).
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data was collected for 1 participant only; and was not presented in order to protect participant confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Invasive Breast Cancer-free Survival (IBCFS)
Description: IBCFS was defined according to standardized definitions for efficacy outcome measure in adjuvant breast cancer trials (STEEP) criteria version 2.0 as the time interval from the date of randomization to the date of the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence (IIBTR): invasive breast cancer involving the same breast parenchyma as the original primary; local-regional invasive breast cancer recurrence: invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast; distant recurrence: metastatic disease-breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer, invasive contralateral breast cancer; death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
Time Frame: From randomization to the date of first occurrence of IBCFS event (maximum exposure duration: 155 days)
Population: No invasive breast cancer event data was collected because of the early termination of the study by the Sponsor and thus IBCFS was not analyzed. Therefore, no data is reported for this outcome measure.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Invasive Disease-Free Survival (IDFS)
Description: IDFS according to STEEP criteria version 2.0 was defined as the time interval from the date of randomization to the date of the first occurrence of one of the following events: IIBTR: invasive breast cancer involving the same breast parenchyma as the original primary; local-regional invasive breast cancer recurrence: invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast; distant recurrence: metastatic disease-breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer; invasive contralateral breast cancer; second non-breast primary invasive cancer; death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
Time Frame: From randomization to the date of first occurrence of IDFS event (maximum exposure duration: 155 days)
Population: No Invasive disease event data was collected because of the early termination of the study by the Sponsor and thus IDFS was not analyzed. Therefore, no data is reported for this outcome measure.
Groups:
- Amcenestrant 200 mg + Tamoxifen-Matching Placebo: Participants received amcenestrant 200 mg along with tamoxifen-matching placebo orally PO, QD from Day 1 to Day 28 of each 28-day treatment cycle and were followed-up until diagnosis of disease recurrence per IBCFS definition included (recurrence of one of following: IIBTR; local-regional invasive breast cancer recurrence; distant recurrence, invasive contralateral breast cancer, death) or any other withdrawal criterion whichever occurs first (maximum exposure duration: 155 days).
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

3. Secondary Outcome: Distant Recurrence-free Survival (DRFS)
Description: DRFS according to STEEP criteria version 2.0 was defined as the time interval from the date of randomization to the date of the first occurrence of one of the following events: distant recurrence or death attributable to any cause (including breast cancer, non-breast cancer, or unknown cause).
Time Frame: From randomization to the date of the first occurrence of distant recurrence or death due to any cause, whichever occurs first (maximum exposure duration: 155 days)
Population: No distant recurrence event data was collected because of the early termination of the study by the Sponsor and thus DRFS was not analyzed. Therefore, no data is reported for this outcome measure.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Locoregional Recurrences-free Survival (LRRFS)
Description: LRRFS was defined as the time interval from the date of randomization to the date of the first occurrence of one of the following events: local/regional ipsilateral recurrence, invasive contralateral breast cancer or death attributable to any cause (including breast cancer, non-breast cancer, or unknown cause).
Time Frame: From randomization to the date of the first occurrence of local/regional ipsilateral recurrence or breast cancer or death due to any cause, whichever occurs first (maximum exposure duration: 155 days)
Population: No locoregional recurrences event data was collected because of the early termination of the study by the Sponsor and thus LRRFS was not analyzed. Therefore, no data is reported for this outcome measure.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time interval from the date of randomization to the date of documented death (due to any cause).
Time Frame: From randomization to the date of death due to any cause (maximum exposure duration: 155 days)
Population: Analysis was performed on randomized population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 3
months | NA [NA to NA] — Median, upper and lower limit of 95% confidence interval (CI) was not estimable as no event was collected.

6. Secondary Outcome: Breast Cancer-specific Survival (BCSS)
Description: BCSS was defined as the time interval from the date of randomization to the date of documented death attributable to breast cancer cause.
Time Frame: From randomization to the date of death due to breast cancer (maximum exposure duration: 155 days)
Population: Analysis was performed on randomized population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 3
months | NA [NA to NA] — Median, upper and lower limit of 95% CI was not estimable as no event was collected.

7. Secondary Outcome: Change From Baseline in Overall Side Effect Bother As Measured By Functional Assessment of Cancer Therapy Item GP-5 (FACT-GP5) Scale Scores
Description: FACT-GP5 is a single-item from the Functional Assessment of Cancer Therapy-General (FACT-G) scale in which participants report their bother by side effects of treatment response. Responses were given on a 5- point Likert-type scale with score range from 0 (not at all bothered by side effect) to 4 (very much bothered by side effects). Higher scores indicate a higher degree of side effect bother. End of treatment (EOT) visit was 30 days after the last IMP administration.
Time Frame: Baseline, Cycle 3, 4, 5, 6, 7, 10, 13, 16, 19, 22, 25, 28, 34, 40, 46, 52, & 58 and at end of treatment (maximum exposure: any day up to 155 days)
Population: Evaluable data was collected for 2 participants only; and thus, was not presented to protect participant confidentiality.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Breast Cancer Specific Module (EORTC-QLQ-BR23): Systemic Therapy Side Effects Scale Score
Description: QLQ-BR23: 23-item disease-specific participant reported outcome measure of disease-related symptoms, treatment-related symptoms, and functioning relevant to participants with breast cancer. It consisted of 4 functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and 4 symptoms scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptom). Systemic therapy side effects scale consisted of 7 items & each item was rated on a 4-point scale with responses as: 1= not at all, 2= a little, 3= quite a bit, 4= very much. A linear transformation was applied to raw scores so that all transformed scores are within 0 to 100. A higher score denotes worse symptoms for the systemic therapy side effects symptom scale. Negative change from baseline= improvement of side effects, positive change = deterioration. EOT visit was 30 days after last IMP administration.
Time Frame: Baseline, Cycle 2, 4, 7, 10, 13, 16, 19, 22, 25, 28, 34, 40, 46, 52, & 58 and at end of treatment (maximum exposure: any day up to 155 days)
Population: Evaluable data was collected for 1 participant only; and was not presented to protect participant confidentiality.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30): Global Health Status/Quality of Life (GHQ) Scale Score
Description: EORTC-QLQ-C30: cancer-specific instrument with 30 questions for evaluation of new chemotherapy & assessment of participant reported outcome. EORTC QLQ-C30 included global health status/quality of life (GHS/QOL), functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from QLQ-C30 were rated on a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were rated on a 7-point scale (1/Very Poor to 7/Excellent). All scales were transformed from raw scores to linear scales ranging 0 to 100. A high score represented a favorable outcome with a best quality of life for participant. EOT visit was 30 days after last IMP administration.
Time Frame: as for outcome 8
Population: Evaluable data was collected for 1 participant only; and was not presented to protect participant confidentiality.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

10. Secondary Outcome: Plasma Concentration of Amcenestrant
Time Frame: Pre-dose on Cycle 2 Day 1, Cycle 7 Day 1, Cycle 13 Day 1 and Cycle 25 Day 1
Population: Data was not collected and analyzed for this outcome measure due to the early termination of the study by the Sponsor.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) data was collected from first dose of study drug administration up to 30 days after the last treatment administration (maximum exposure duration:155 days)
Description: Analysis was performed on all randomized population.
Arm/Group | Amcenestrant 200 mg + Tamoxifen-Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amcenestrant 200 mg + Tamoxifen-Matching Placebo (N=3)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Glucose Intolerance (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to premature discontinuation and closure of study decided by the Sponsor, only safety data were summarized and reported, and no efficacy data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT05128773/Prot_SAP_000.pdf